CLINICAL TRIAL: NCT03473795
Title: Developing Non-Communicable Disease Registries in Africa: A Step Towards Providing Quality Data for Improving Patient Outcomes
Brief Title: Developing Non-Communicable Disease Registries in Africa : A Step Towards Providing Quality Data for Improving Patient Outcomes
Status: Enrolling by invitation | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Duke University (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: 18-114
Record Dates: First submitted 2018-03-16; First posted 2018-03-22 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Non-Communicable Disease
Keywords: Patient Outcomes; 18-114
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Samples can include tissue, blood, urine, saliva, hair and nail clipping.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy participants and participants diagnosed with NCDs: This protocol will entail prospective collection of data on healthy participants and participants diagnosed with NCDs managed at collaborating institutions in SSA. Information to be obtained includes socio-demographic data, risk factors, disease-specific data, investigation and treatment details, as well as findings during follow-up. Particular reference will be made to outcome measures such as local and distant recurrence, survival and mortality. Follow-up data will be updated during clinic visits and also via phone calls.
  Interventions: Behavioral: Questionnaire forms; Other: Bio-specimen samples

INTERVENTIONS:
Behavioral: Questionnaire forms — The questionnaires will include information such as socio-demographic data, risk factors, disease specific data, investigation and treatment details as well as findings during followup. Particular reference will be made to outcome measures such as local and distant recurrence, survival and mortality.
Other: Bio-specimen samples — Samples can include tissue, blood, urine, saliva, hair and nail clipping.

SUMMARY:
This umbrella protocol seeks to develop robust data registries for non-communicable diseases (NCDs) in sub-Saharan Africa (SSA) with the aim of providing accurate and comprehensive data for the evaluation of such diseases in sub-Saharan African countries.Healthy volunteers will be included in the study for comparison.

Additionally, the investigators aim to describe the gut microbiome community diversity of a cohort of community dwelling Nigerians and compare with CRC patients in Nigerian and at MSK. We will collect stool for microbiome and metabolomic analysis from community dwelling persons in the catchment area of ARGO facilities in Nigeria while contemporaneously administering an extensive medical and environmental exposure questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older.
* Suspected or confirmed diagnosis of a non-communicable disease. OR
* Healthy volunteers/no confirmed diagnosis for comparison.

Exclusion Criteria:

* Participants unwilling to sign consent.
* Participants under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be accrued in medical clinics in Africa as determined by the local investigators and local research staff.
Sampling Method: Non-Probability Sample
Enrollment: 7566 (Estimated)
Dates: Start 2018-03-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
# of patients that develope non-communicable diseases in Africa | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: T. Peter Kingham, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (14):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States
- Nigeria (13):
  - National Hospital of Abuja (Data collection only), Abuja, Central Business District
  - Lagos State University Teaching Hospital, Idi Araba, Lagos
  - Olabisis Onabanjo University Teaching Hospital, Sagamu, Ogun State
  - Federal Medical Centre Owo, Owo, Ondo State
  - University College Hospital, Ibadan, Oyo State
  - Ladoke Akintola University of Technology, Ogbomoso, Oyo State
  - University Of Nigeria Teaching Hospital (UNTH) Ituku-Ozalla Enugu, Enugu
  - Lagos State University Teaching Hospital, Ikeja
  - Obafemi Awolowo University Teaching Hospitals Complex (OAUTHC), Ile-Ife
  - University of Ilorin Teaching Hospitals, Ilorin
  - University of Maiduguri Teaching Hospital (Data collection only), Maiduguri
  - Ondo State Trauma and Surgical Centre, Ondo
  - Federal Medical Centre Owo, Owo

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm